CLINICAL TRIAL: NCT04726163
Title: Tele-expertise for Glycemic Control Monitoring in Patients With Diabetes Hospitalized for Covid-19 Infection
Brief Title: Tele-expertise in Patients With Diabetes Hospitalized for Covid-19 Infection
Acronym: COVIDEX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inclusion difficulties
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 8078
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Diabetic Patient (Type 1,2, MODY, Secondary) or With Corticosteroid-induced Diabetes Following Initiation of Corticosteroid Treatment
Keywords: Diabetes; Covid-19; Telemedecine; Continuous glucose monitoring; Steroid therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Neoplasm Metastasis; Diabetes Mellitus; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-expertise (No Intervention): Basal-bolus insulin treatment with adaptation of insulin doses according to continuous glucose measurement
- Standard (Experimental): Standard treatment and adaptation of insulin doses according to the usual management of the unit
  Interventions: Device: Continuous blind glucose measurement device (Free style Pro)

INTERVENTIONS:
Device: Continuous blind glucose measurement device (Free style Pro) — A continuous blind glucose measurement device (Free style Pro) will be set up on the first day and throughout the entire hospital stay
  Arms: Standard

SUMMARY:
Diabetes is a major factor of morbi-mortality in Covid-19 infection. Currently, steroid therapy is required in patients under oxygen therapy. This treatment is associated with hyper glycaemia in patients with diabetes. Recommendations for the management of diabetes during Covid-19 infection is to use insulin treatment. The majority of units involves in the management of patient with Covid19 infection are not the experience in managing intensive insulin therapy and the time to ensure this follow-up. All the data in the literature are in favor of a positive impact of telemedicine on the metabolic control of diabetic patients. However, the routine use of telemedicine and more particularly tele-expertise within hospital units is very underdeveloped in France. The epidemic of Covid-19 represents a unique situation where the health authorities recommend to physicians to use telemedicine to ensure the follow-up and optimal management of patients. The aim of this study was to compare the metabolic control of diabetic patients infected with Covid-19 followed in tele-expertise to a group of diabetic patients infected with Covid-19 managed in standard conditions.

DETAILED DESCRIPTION:
The study will take place in the infectious diseases department of the University Hospitals of Strasbourg. All diabetic patients or patients with corticosteroid-induced diabetes hospitalized for Covid-19 infection and requiring corticosteroid therapy (Dexamethasone 6mg / day IV for 10 days or Solupred 40mg / day per os) can be recruited.

Subjects meeting the eligibility criteria will be informed of the research orally and by the delivery of a written information notice from the start of their hospitalization in the department:

The allocation of the study group will be made according to the patient's hospitalization unit in the infectious disease department, unit 1 will benefit from tele-expertise (TE group) and patients in unit 2 will belong to the standard group (group S). Unit 1 and Unit 2 of the infectious disease department take care of patients in the same way..

The TE group consists of patients treated from the start of steroid therapy with a basal / bolus insulin regimen at a dose of 0.5U / kg / day: 50% in basal insulin Abasaglar and 50% in rapid insulin Humalog divided into three prandial injections with adaptation of insulin doses on the basis of the MCG. The use of the MCG with a collection of 90 glycemia / day allows the establishment of an intensive insulin treatment in complete safety because of the access to postprandial glycemia for the adaptation of rapid insulin and glycemia nocturnal for adaptation of basal insulin. The implementation of a basal bolus insulin therapy in a non-diabetes unit is made possible by continuous glucose measurement. Freestyle libre will therefore be implemented as soon as the insulin treatment is carried out. The Freestyle libre continuous glucose measurement sensor provides access to 90 interstitial glucose measurements / day and the establishment of continuous glucose measurement curves sent by secure computer every 48 hours for diabetes advice and dose adjustment insulin It is suggested for the study to carry out at least 8 glucose measurements / day per Free style Libre scanner. Therefore, there will be no achievement of capillary blood glucose in the TE group

The standard group (S) consists of patients for whom diabetes management is carried out according to the habits of the infectious disease department. This standard care includes the initiation of insulin therapy (one to several injections of insulin per day) in a context of hyperglycemia according to the habits of the department. The adjustment of the insulin doses in the S group will be carried out on the basis of at least 3 capillary blood glucose tests per day carried out before each meal. Group S will benefit from the fitting of a Freestyle Libre Pro, that is to say a continuous glucose sensor fitted throughout the hospital stay. The Freestyle Libre Pro, does not provide access to real-time interstitial glucose readings but has the option once removed to be able to analyze all 90 interstitial glucose readings. Its interest is to avoid interfering with the standard diabetes management of the infectious disease department.

ELIGIBILITY:
Inclusion Criteria:

* Patient adult hospitalized for Covid-19 infection in the Infectious Diseases Department of the University Hospital of Strasbourg (HUS)
* Patient requiring steroid treatment
* Diabetic patient (type 1,2, MODY, secondary) or with corticosteroid-induced diabetes following initiation of corticosteroid treatment

Exclusion Criteria:

* Contraindication to the use of the Free-Style Medical Device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent in the range 70-180 mg / dl (TIR) | At the end of hospitalization (maximum day 14)
  measured every day in the group followed by tele-expertise compared with group under standard care (comparison of the daily evolution of the TIR in both groups).

SECONDARY OUTCOMES:
Mortality | At the end of hospitalization (maximum day 14)
Intensive Care Unit Transfers | At the end of hospitalization (maximum day 14)
Cardiovascular and infectious complications | At the end of hospitalization (maximum day 14)
Acute metabolic complications: keto acidosis, severe hypoglycaemia | At the end of hospitalization (maximum day 14)
Duration of hospitalization and treatments administered | At the end of hospitalization (maximum day 14)
Mean glucose | At the end of hospitalization (maximum day 14)
Time spent above glycaemia > 180mg/dl | At the end of hospitalization (maximum day 14)
Time spent bellow glycaemia < 70mg/dl | At the end of hospitalization (maximum day 14)

CONTACTS AND LOCATIONS:
Locations (1):
- Hopitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided